CLINICAL TRIAL: NCT00861471
Title: Phase I/II, Open Label Study of Sequential Taxotere® (Docetaxel) and Gleevec® (Imatinib Mesylate) in Hormone Refractory Prostate Cancer
Brief Title: Docetaxel (Taxotere) and Imatinib Mesylate (Gleevec) in Hormone Refractory Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: due to slow accrual
Sponsor: NYU Langone Health (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYU 04-47 (H12554); Novartis CSTI571BUS200 (Other: Novartis)
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Results first posted 2011-06-29 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-05

CONDITIONS: Prostate Cancer; Prostatic Neoplasms
Keywords: hormone refractory prostate cancer; tyrosine kinase inhibitor; Gleevec; PSA; prostate specific antigen; growth factor receptor inhibitor; androgen independent
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel +Gleevec (Experimental)
  Interventions: Drug: Docetaxel; Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Docetaxel — One treatment cycle is defined as 21 days.
  Docetaxel: 70 mg/m^2 (60 mg/m^2 was tested in Phase I as well), Intravenous, every 21 days.
  Other Names: Taxotere
Drug: Imatinib Mesylate — One treatment cycle is defined as 21 days.
  Imatinib Mesylate: 24-36 hours after Docetaxel, 600 mg (400 mg was tested in Phase I as well), orally, daily x 14 days.
  Other Names: Gleevec

SUMMARY:
This trial is designed to determine the proper doses of Docetaxel and Imatinib mesylate to be used to treat hormone refractory prostate cancer and to evaluate the safety and efficacy of the treatment.

DETAILED DESCRIPTION:
Androgen-independent prostate cancer is the second most common cause of cancer death in men. These patients have limited treatment options. Docetaxel(Taxotere) is the single most active agent for the treatment of hormone refractory prostate cancer. Phase II clinical trials including docetaxel combinations with other microtubule inhibitors have shown 60-70% prostate specific antigen (PSA) declines greater than 50% and 30-40% measurable disease responses. However, the duration of response is limited to roughly 22 weeks. Combinations with new agents are needed to increase the rate and duration of response over existing docetaxel containing combinations.

The platelet derived growth factor receptor(PDGFR)and platelet derived growth factor (PDGF) A are frequently expressed (80%) in primary and bone marrow metastasis of human prostate cancer (PC). Recent experimental evidence suggests that activation of PDGFR/PDGF can be oncogenic in the development and/or progression of PC. There is also evidence that PC cells that express PDGF promote PDGFR expression in endothelial cells and neo- angiogenesis. Together, these experimental evidence supports that inhibition of PDGFR may be of therapeutic benefit to advanced prostate cancer patients.

Gleevec (Imatinib mesylate ) is a potent inhibitor of PDGFR. Consistent with these observations, treatment with Gleevec in an experimental prostate cancer mouse model was better than paclitaxel alone in reducing bone metastasis but the antitumor effect was strongest with the combination of both. In a phase I study of heavily pretreated hormone refractory PC patients, Gleevec 600 mg/daily lead-in for 30 days followed by Gleevec 600 mg/daily with Paclitaxel 30mg/m2 weekly x4 weeks every 6 weeks induced a >50% PSA decline in 7% and 38% of patients respectively with acceptable toxicity. These observations suggested that this combination merits further investigation.

With high-dose docetaxel (70mg/m^2) being the single most active agent in hormone refractory prostate cancer and no data existing in the use of high-docetaxel with Gleevec, a phase I/II study to determine the maximum tolerated dose (MTD) of the combination and optimum dose for a phase II trial is warranted.

Gleevec is expected to affect the activation status of sensitive receptor tyrosine kinase targets and associated signaling effectors in the tumor cells and the neovasculature. However, it is not fully established to what extent alterations of the target and /or other molecules in the signaling pathway are essential for Gleevec's antitumor activity in prostate cancer patients. It is also unknown whether preexisting molecular changes in the prostate tumors of individual patients could affect Gleevec's activity even in the presence of the targets. Therefore, an assessment of the expression levels and/or presence of mutations of selected molecules in specimens of patients in clinical trials may contribute in various ways: 1. to understand the requirements to elicit or inhibit a response to the combination, 2. whether adding other targeted agents may improve response and/or 3. whether selection of patients that might benefit should be based on the tumor profile. Thus, whenever possible specimens form the primary and/or metastatic sites should be retrieved and/or obtained to perform these analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age.
* Histologically documented diagnosis of adenocarcinoma of prostate gland
* Patients must have hormone refractory prostate cancer having progressed after at least two prior hormonal manipulations with documented castrate levels of testosterone (<50 ng/dl). PSA ≥ 5 ng/ml
* Patients must have hormone-refractory prostate carcinoma as evidenced by PSA progression, with or without evidence of measurable disease, or evaluable disease by a positive bone scan. PSA progression is defined as > 25% increase in 2 consecutive tests in which the first increase in PSA should occur a minimum of 1 week from the reference value and this increase in PSA should be confirmed and ≥ 5 ng/ml
* Eligible patients will have been treated with at least two prior hormonal manipulations including androgen deprivation and may have received one prior chemotherapy regimen.
* Any chemotherapy, major surgery, or irradiation must have been completed at least 3 weeks prior to starting study drugs. Patient must have recovered from clinically significant toxicities incurred as a result of previous therapy except nail dystrophy, alopecia, grade 1 peripheral neuropathy, or radiation therapy induced affects (i.e., impotence or incontinence)
* No recent prior flutamide (Eulexin) use within the past 4 weeks, prior bicalutamide (Casodex) use within the past 6 weeks, or prior nilutamide (Nilandron) use within the past 6 weeks.
* Performance status 0,1, 2 (Eastern Cooperative Oncology Group performance status scale)
* Adequate end organ function, defined as the following:

  * total bilirubin < 1.5 x upper limit of Normal (ULN)
  * Serum glutamic-oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) < 2.5 x ULN
  * creatinine < 1.5 x ULN
  * Absolute Neutrophil count (ANC) > 1.5 x 10^9/L
  * platelets > 100 x 10^9/L
* Written, voluntary informed consent.
* Patients must have been and continue to be on androgen deprivation therapy with a Luteinizing hormone-releasing hormone (LHRH) agonist or antagonist during study participation except for patients who had orchiectomy.
* Patients on secondary hormonal manipulation with ketoconazole and hydrocortisone who discontinued LHRH therapy must be switched to single agent LHRH analogue therapy unless they had orchiectomy.
* Patients being treated with Zometa prior to the initiation of the study will be permitted to continue with Zometa while on the study.

Exclusion Criteria:

* Patient has received any other investigational agents within 28 days of first day of study drug dosing, unless the disease is rapidly progressing.
* Patient is < 5 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
* Patient with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months of study)
* Patient has a severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection).
* Patient with untreated brain metastasis or cord compression. However, patients with treated spinal cord compression or central nervous system (CNS) metastases that have been stable are eligible.
* Patient has known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
* Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
* Patient received chemotherapy within 4 weeks (6 weeks for nitrosourea or mitomycin-C) prior to study entry, unless the disease is rapidly progressing.
* Patient previously received radiotherapy to at least 25 % of the bone marrow
* Patient had a major surgery within 2 weeks prior to study entry.
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.
* If the patient is taking steroids for prostate cancer, then the patient is ineligible for this study. If the patient is taking steroids for conditions other than prostate cancer, the patient is eligible provided that the reasons for use and dosage are documented. The investigator is urged to discuss this issue with the Study Principal Investigator for any clarification.
* No therapeutic anticoagulation with warfarin (e.g. Coumadin® or Coumadine®) will be permitted in patients participating in this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Ferrari, MD, Principal Investigator — New York University Cancer Institute
Locations (3):
- United States (3):
  - Bellevue Hospital, New York, New York
  - NYU Clinical Cancer Center, New York, New York
  - NYU Tisch Hospital, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 patients were enrolled between Sep. 2006 and Nov. 2008 for the Phase II part of the study in New York University Medical center and affiliated hospitals.
Pre-assignment Details: Once the optimal combination dose of Docetaxel (Taxotere) and Gleevec (Imatinib Mesylate) was determined in the Phase I part, the study proceeded to Phase II. There were 12 patients in Phase I and Phase II, respectively. The results reported here are only for Phase II.
Groups:
- Docetaxel +Gleevec: 21 days per treatment cycle for up to 1 year: Day 1: Docetaxel (Taxotere) ( 70 mg/m^2 intravenously over 1 hour. Day 2: (24-36 hours later) start Gleevec (Imatinib Mesylate) 600 mg, orally, daily x 14 days
Period: Overall Study
Arm/Group | Docetaxel +Gleevec
Started | 12
Completed | 3
Not Completed | 9
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 3
Not completed — treatment for lumbar laminectomy | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel +Gleevec
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Prostate Specific Antigen (PSA) Response
Description: PSA response is defined as a greater than or equal to a 50% decrease in PSA from the baseline without clinical or radiologic evidence of progression according to the Response Evaluation Criteria in Solid Tumors (RECIST). PSA concentration was measured at baseline on day 1/cycle 1 before treatment, then day 1 of every cycle afterwards during therapy.
Time Frame: up to 9 months
Population: The analysis was based on intent-to-treat population.
Measure: Number; unit: percentage of participants
Arm/Group | Docetaxel +Gleevec
Number analyzed (Participants) | 12
percentage of participants | 50

2. Secondary Outcome: Percentage of Participants With Greater or Equal to 80% PSA Reduction From Baseline Without Clinical or Radiologic Evidence of Progression
Description: PSA was measured at baseline on day 1/cycle 1 before treatment, then day 1 of every cycle afterwards during therapy.
Time Frame: up to 9 months
Population: The analysis was based on intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Docetaxel +Gleevec
Number analyzed (Participants) | 12
percentage of participants | 16

3. Secondary Outcome: Percentage of Participants With Measurable Disease Response
Description: Measurable disease response is defined as the number of participants whose best response is complete response or partial response over the number of patients with measurable desease according to the Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: up to 2 years
Population: Based on the participants with measurable disease
Measure: Number; unit: percentage of participants
Arm/Group | Docetaxel +Gleevec
Number analyzed (Participants) | 5
percentage of participants | 20

4. Secondary Outcome: Time to PSA Progression
Description: Time to PSA pregression is defined as the time at which therapy statred and ends when the PSA increased by 50% above the nadir confirmed on a second determination.
Time Frame: up to 2 years
Population: Based on intent-to-treat population
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Docetaxel +Gleevec
Number analyzed (Participants) | 12
days | 188 [85 to 279]

5. Secondary Outcome: Median Overall Survival Time
Description: Overall survival time is the time from the start of therapy till death. Median overall survival reported here is the time when 50% of the participants are alive.
Time Frame: up to 4 years
Population: Based on intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel +Gleevec
Number analyzed (Participants) | 12
months | 24.9 [14.3 to 35.4]

ADVERSE EVENTS:
Time Frame: on study (up to 9 months) plus 30 days after
Description: adverse events were collected by patient reporting, investigator questioning, physical exams, lab tests, etc.
Arm/Group | Docetaxel +Gleevec
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel +Gleevec (N=12)
Sinus tachycardia (Cardiac disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
infection with normal ANC (Infections and infestations) | 1 (1)
pain-other (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel +Gleevec (N=12)
abdominal pain or cramping (General disorders) | 2
allergic rhinitis (Immune system disorders) | 1
alopecia (Skin and subcutaneous tissue disorders) | 5
anorexia (Gastrointestinal disorders) | 4
bone pain (Musculoskeletal and connective tissue disorders) | 1
constipation (Gastrointestinal disorders) | 4
constitutioanl symptoms-other (General disorders) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 2
dehydration (Gastrointestinal disorders) | 1
dermotology/ skin- other (Skin and subcutaneous tissue disorders) | 4
diarrhea (with colostomy) (Gastrointestinal disorders) | 1
diarrhea (without colostomy) (Gastrointestinal disorders) | 5
dry skin (Skin and subcutaneous tissue disorders) | 2
dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
edema (Cardiac disorders) | 5
fatigue (General disorders) | 9
fever (General disorders) | 1
gastrointestinal- other (Gastrointestinal disorders) | 1
hemoglobin (Blood and lymphatic system disorders) | 8
hyponatremia (Metabolism and nutrition disorders) | 1
injection site reaction (Skin and subcutaneous tissue disorders) | 1
insomnia (Nervous system disorders) | 1
leukocytes (Blood and lymphatic system disorders) | 1
lymphatics (Blood and lymphatic system disorders) | 3
myalgia (Musculoskeletal and connective tissue disorders) | 2
nail changes (Skin and subcutaneous tissue disorders) | 4
nausea (Gastrointestinal disorders) | 7
neuropathy /sensory (Nervous system disorders) | 7
neutrophils/ granulocytes (Blood and lymphatic system disorders) | 2
ocular/ visual -other (Eye disorders) | 3
pain -other (General disorders) | 3
palpitations (Cardiac disorders) | 1
platelets (Blood and lymphatic system disorders) | 1
pruritus (Skin and subcutaneous tissue disorders) | 1
rash/ desquamation (Skin and subcutaneous tissue disorders) | 1
rigors/ chills (General disorders) | 1
sinus tachycardia (Cardiac disorders) | 1
stomatitis/ pharyngitis (Gastrointestinal disorders) | 1
taste disturbance (Gastrointestinal disorders) | 4
tearing (Eye disorders) | 3
vomiting (Gastrointestinal disorders) | 3
weight gain (General disorders) | 1
weight loss (General disorders) | 1

LIMITATIONS AND CAVEATS:
This study was terminated before it reached the target accrual number due to slow accrual, leading to small number of subjects analyzed (12 out of the target number of 37).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes